CLINICAL TRIAL: NCT02249832
Title: The General Use of Robots in Stroke Recovery: the Anklebot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Bruce Volpe, Principal Investigator, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-310
Record Dates: First submitted 2014-09-23; First posted 2014-09-26 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2021-03-09 (Actual); Status verified 2019-11

CONDITIONS: Stroke
Keywords: stroke; CVA; cerebrovascular accident; cerebral stroke; robotic therapy; anklebot; physical therapy
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Intervention Model Description: All subjects received 18 sessions (3 times per week for 6 weeks) of seated robotic ankle training. Upon analysis, subjects were stratified by average admission gait speed on the 10 Meter Walk Test at comfortable pace, according to clinically established gait speed performance groups: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) gait functioning.
Oversight: Data Monitoring Committee: No

ARMS (1):
- seated robot-assisted ankle therapy (Experimental): All participants received eighteen 1 hour sessions (3x/week for 6 weeks) of seated robot-assisted ankle training with the MIT anklebot. Upon analysis, subjects were stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to clinically established gait speed performance groups: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) functioning.
  Interventions: Device: seated robot-assisted ankle therapy

INTERVENTIONS:
Device: seated robot-assisted ankle therapy — The MIT anklebot provides over one thousand total dorsi/plantar flexion and inversion/eversion robot-assisted movements of the ankle while in a seated position.
  Other Names: Massachusetts Insititute of Technology (MIT) Anklebot

SUMMARY:
The purpose of this study is to determine if isolated robot-assisted training of the ankle joint improves chronic hemiparetic gait in patients after stroke.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* First single focal unilateral lesion with diagnosis verified by brain imaging, which occurred at least 6 months prior
* Cognitive function sufficient enough to understand experiments and follow instructions
* Some amount of independent ambulation (with orthoses or walker)

Exclusion Criteria:

* Botox treatment within 6-weeks of enrollment;
* Fixed contraction deformity in the affected limb;
* Complete and total flaccid paralysis of all lower extremity motor function;
* Unable to ambulate except with the aid of another person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2013-06; Primary Completion 2019-02 (Actual); Study Completion 2019-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Feinstein Institutes for Medical Research, Manhasset, New York
  - Transitions of Long Island Outpatient Rehabilitation, Manhasset, New York

REFERENCES:
- [Background] Khanna I, Roy A, Rodgers MM, Krebs HI, Macko RM, Forrester LW. Effects of unilateral robotic limb loading on gait characteristics in subjects with chronic stroke. J Neuroeng Rehabil. 2010 May 21;7:23. doi: 10.1186/1743-0003-7-23. PMID 20492698
- [Background] Roy A, Krebs HI, Bever CT, Forrester LW, Macko RF, Hogan N. Measurement of passive ankle stiffness in subjects with chronic hemiparesis using a novel ankle robot. J Neurophysiol. 2011 May;105(5):2132-49. doi: 10.1152/jn.01014.2010. Epub 2011 Feb 23. PMID 21346215
- [Background] Forrester LW, Roy A, Krebs HI, Macko RF. Ankle training with a robotic device improves hemiparetic gait after a stroke. Neurorehabil Neural Repair. 2011 May;25(4):369-77. doi: 10.1177/1545968310388291. Epub 2010 Nov 29. PMID 21115945
- [Background] Forrester LW, Roy A, Krywonis A, Kehs G, Krebs HI, Macko RF. Modular ankle robotics training in early subacute stroke: a randomized controlled pilot study. Neurorehabil Neural Repair. 2014 Sep;28(7):678-87. doi: 10.1177/1545968314521004. Epub 2014 Feb 10. PMID 24515923

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants received eighteen sessions of seated anklebot training. Upon analysis, subjects were stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to well standardized gait speed performance groups: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) functioning.
Groups:
- Seated Robotic Ankle Therapy: Participants received eighteen 1 hour sessions (3 times/week for 6 weeks) of seated anklebot training with the MIT Anklebot.
Period: Overall Study
Arm/Group | Seated Robotic Ankle Therapy
Started | 55
Completed | 42
Not Completed | 13
Not completed — Withdrawal by Subject | 3
Not completed — Lost to Follow-up | 10

BASELINE CHARACTERISTICS:
Groups:
- Seated Robotic Ankle Therapy: Participants received eighteen, 1 hour sessions (3 times/week for 6 weeks) of seated anklebot training with the MIT Anklebot.
Arm/Group | Seated Robotic Ankle Therapy
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 40
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Gait Speed (m/Sec) on the 10 Meter Walk Test at Comfortable Pace.
Description: Subjects were stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to clinically established gait speed performance groups: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) functioning. Mean gait speeds on the 10m Walk Test at comfortable pace (m/sec) were then compared across these three groups (low, moderate, and high function) at three timepoints (baseline, discharge (week 6), and 3 month FU (overall week 18)).
Time Frame: baseline, discharge (week 6), 3 month FU (overall week 18)
Population: Subjects were stratified according to clinically established gait speed impairment levels based on average admission gait speed on the 10 Meter Walk Test at comfortable pace.
Measure: Mean (Standard Error); unit: m/sec
Groups:
- Low Gait Speed Group: The low gait speed group included all subjects with a mean gait speed of <0.4m/sec on the admission 10 Meter Walk Test at comfortable pace, based upon clinically established gait speed performance levels.
- Moderate Gait Speed Group: The moderate gait speed group included all subjects with a mean gait speed of 0.4-0.8m/sec on the admission 10 Meter Walk Test at comfortable pace, based upon clinically established gait speed performance levels.
- High Gait Speed Group: The high gait speed group included all subjects with a mean gait speed of >0.8m/sec on the admission 10 Meter Walk Test at comfortable pace, based upon clinically established gait speed performance levels.
Arm/Group | Low Gait Speed Group | Moderate Gait Speed Group | High Gait Speed Group
Number analyzed (Participants) | 21 | 14 | 7
m/sec
  Mean gait speed at baseline | 0.22 (0.02) | 0.53 (0.03) | 1.02 (0.07)
  Mean gait speed at discharge (week 6) | 0.26 (0.02) | 0.62 (0.04) | 1.18 (0.12)
  Mean gait speed at 3month FU (overall week 18) | 0.24 (0.02) | 0.66 (0.04) | 1.29 (0.10)
Statistical Analysis 1: Comparison: Low Gait Speed Group vs Moderate Gait Speed Group vs High Gait Speed Group; Test type: Equivalence — A 3x3 repeated measures ANOVA was performed with group (mean gait speed in the low, moderate, and high groups) and time (admission, discharge (week 6), and follow-up (overall week 18) in each condition) as factors. Null hypothesis was that there was no difference in mean gait speed over time across the three groups. A significance level of 0.05 was used (two-sided); p < 0.001, ANOVA — A significance level of 0.05 was used (two-sided)

2. Secondary Outcome: Mean Change From Baseline in Gait Speed (m/Sec) on the 10 Meter Walk Test at Fast Pace.
Description: Subjects were stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to clinically established gait speed performance groups: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) functioning. Mean gait speeds on the 10m Walk Test at fast pace (m/sec) were then compared across these three groups (low, moderate, and high function) at three timepoints (baseline, discharge (week 6), and 3 month FU (overall week 18)).
Time Frame: baseline, discharge (week 6), 3 month FU (overall week 18)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: m/sec
Groups:
- Low Gait Speed Group: The low gait speed group included all subjects with a mean gait speed of <0.4m/sec on the admission 10 Meter Walk Test at comfortable pace, based upon clinically established gait speed impairment levels.
- Moderate Gait Speed Group: The moderate gait speed group included all subjects with a mean gait speed of 0.4-0.8m/sec on the admission 10 Meter Walk Test at comfortable pace, based upon clinically established gait speed impairment levels.
- High Gait Speed Group: The high gait speed group included all subjects with a mean gait speed of >0.8m/sec on the admission 10 Meter Walk Test at comfortable pace, based upon clinically established gait speed impairment levels.
Arm/Group | Low Gait Speed Group | Moderate Gait Speed Group | High Gait Speed Group
Number analyzed (Participants) | 21 | 14 | 7
m/sec
  mean gait speed at baseline | 0.25 (0.02) | 0.67 (0.06) | 1.30 (0.13)
  mean gait speed at discharge (week 6) | 0.29 (0.03) | 0.79 (0.06) | 1.41 (0.18)
  mean gait speed at 3 month FU (overall week 18) | 0.27 (0.03) | 0.84 (0.10) | 1.79 (0.26)
Statistical Analysis 1: Comparison: Low Gait Speed Group vs Moderate Gait Speed Group vs High Gait Speed Group; A 3x3 repeated measures ANOVA was performed with group (mean gait speed in the low, moderate, and high groups) and time (admission, discharge (week 6), and follow-up (overall week 18) in each condition) as factors. Null hypothesis was that there was no difference in mean gait speed over time across the three groups. A significance level of 0.05 was used (two-sided); Test type: Equivalence — A significance level of 0.05 was used (two-sided); p < 0.001, ANOVA

3. Secondary Outcome: Mean Change From Baseline in Distance Walked (Meters) on the 6 Minute Walk Test at Comfortable Pace.
Description: Subjects were stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to clinically established gait speed performance groups: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) functioning. Mean distance walked (m) on the 6 Minute Walk test at comfortable pace were then compared across these three groups (low, moderate, and high function) at three timepoints (baseline, discharge (week 6), and 3 month FU (overall week 18)).
Time Frame: baseline, discharge (week 6), 3 month FU (overall week 18)
Population: Subjects were stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to clinically established gait speed performance levels.
Measure: Mean (Standard Error); unit: meters
Arm/Group | Low Gait Speed Group | Moderate Gait Speed Group | High Gait Speed Group
Number analyzed (Participants) | 21 | 14 | 7
meters
  mean distance at baseline | 68.46 (5.76) | 152.92 (9.53) | 280.43 (19.19)
  mean distance at discharge (week 6) | 79.33 (5.38) | 180.11 (11.64) | 319.79 (22.91)
  mean distance at 3 month FU (overall week18) | 75.07 (5.62) | 183.34 (14.33) | 314.43 (21.46)
Statistical Analysis 1: Comparison: Low Gait Speed Group vs Moderate Gait Speed Group vs High Gait Speed Group; Test type: Equivalence — A 3x3 repeated measures ANOVA was performed with group (mean distance walked in the low, moderate, and high groups) and time (admission, discharge (week 6), and follow-up (overall week 18) in each condition) as factors. Null hypothesis was that there was no difference in mean gait speed over time across the three groups. A significance level of 0.05 was used (two-sided); p = 0.001, ANOVA — A significance level of 0.05 was used (two-sided)

ADVERSE EVENTS:
Time Frame: eighteen weeks for each subject (6 weeks of ankle training + 12 week FU period).
Description: Safety population included all participants who enrolled in the study.
Groups:
- Seated Robotic Ankle Therapy: All participants received eighteen 1 hour sessions (3x/week for 6 weeks) of seated anklebot training with the MIT anklebot. Prior to the intervention, subjects were initially stratified based on average admission gait speed on the 10 Meter Walk Test at comfortable pace according to well standardized and accepted gait speed performance levels: low (<0.4m/sec), moderate (0.4m/sec-0.8m/sec) and high (>0.8m/sec) functioning, in order to determine if there were impairment-level differences in the recovery pattern following ankle training.
Arm/Group | Seated Robotic Ankle Therapy
All-Cause Mortality (participants affected / at risk) | 0/55
Serious Adverse Events (participants affected / at risk) | 1/55
Other Adverse Events (participants affected / at risk) | 2/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seated Robotic Ankle Therapy (N=55)
worsening baseline ankle pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Seated Robotic Ankle Therapy (N=55)
neuropathic pain (Nervous system disorders) | 1 (1)
depression (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT02249832/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-31): https://cdn.clinicaltrials.gov/large-docs/32/NCT02249832/ICF_001.pdf